CLINICAL TRIAL: NCT00271830
Title: Sexual Function in Male Renal Transplant Patients
Status: Terminated | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Other Study IDs: MMCIRB05-07-184
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Renal Transplant Recipients
Keywords: renal; transplant; sexual dysfunction; male; dialysis free
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Sexual dysfunction is common in male patients with chronic renal failure on dialysis and after renal trasnplantation. Multiple factors play a role in this important clinical problem. Recent studies suggest that certain immunosuppressive medication used for solid organ transplant may affect male sexual function. The purpose of this study is to compare the sexual function of male renal transplant patients on sirolimus and those patients not on sirolimus immunosuppression.

DETAILED DESCRIPTION:
All male renal transplant recipients with a functioning allograft 1 month post transplant will be eligible to participate in this prospective serial observation study. As roughly half of renal transplant patients are assigned to rapamycin immunnosuppression clinically and half are not, we plan to assess routine clinical perameters, sex hormone levels, subjective sexual function as measured by standardized questionnaire and semen analysis in 55 patients on sirolimus treatment and 55 patients not on this treatment. Assessment will be made at baseline (1 mo post transplant) and 6 and 12 months later. All adult male renal transplant recipients ages 21-65 off dialysis 1 mo post transplant will be eleigible. Exclusion criteria will be female gender, patients requiring testosterone therapy, patients on dialysis, and those unwilling to give informed consent.

ELIGIBILITY:
Inclusion Criteria:male renal transplant recipients off dialysis by 1 month post transplant, ages 21-65,willing to give informed consent

-

Exclusion Criteria: female gender, patients requiring testosterone replacement treatment, patients with neglibile renal function requiring dialysis, unwilling to give informed consent

-

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2006-01; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Glicklich, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States